CLINICAL TRIAL: NCT03739866
Title: A Phase 1b Randomized, Double-Blinded, Placebo Controlled, Multi-Cohort Study of the Safety, Pharmacokinetics, and Antiviral Activity of GS-6207 Administered Subcutaneously in HIV-1 Infected Subjects
Brief Title: Study to Evaluate Safety, Pharmacokinetics, and Antiviral Activity of Lenacapavir Administered Subcutaneously in Human Immunodeficiency Virus (HIV) -1 Infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-200-4072
Record Dates: First submitted 2018-11-02; First posted 2018-11-14 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — lenacapavir; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: Lenacapavir 20 mg (Experimental): Participants will receive single dose of lenacapavir 20 mg on Day 1 followed by bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) as per standard-care therapy starting on Day 10 through Day 225.
  Interventions: Drug: Lenacapavir; Drug: B/F/TAF
- Part A: Lenacapavir 50 mg (Experimental): Participants will receive single dose of lenacapavir 50 mg on Day 1 followed by B/F/TAF as per standard-care therapy starting on Day 10 through Day 225.
  Interventions: Drug: Lenacapavir; Drug: B/F/TAF
- Part A: Lenacapavir 150 mg (Experimental): Participants will receive single dose of lenacapavir 150 mg on Day 1 followed by B/F/TAF as per standard-care therapy starting on Day 10 through Day 225.
  Interventions: Drug: Lenacapavir; Drug: B/F/TAF
- Part A: Lenacapavir 450 mg (Experimental): Participants will receive single dose of lenacapavir 450 mg on Day 1 followed by B/F/TAF as per standard-care therapy starting on Day 10 through Day 225.
  Interventions: Drug: Lenacapavir; Drug: B/F/TAF
- Part A: Lenacapavir 750 mg (Experimental): Participants will receive single dose of lenacapavir 750 mg on Day 1 followed by B/F/TAF as per standard-care therapy starting on Day 10 through Day 225.
  Interventions: Drug: Lenacapavir; Drug: B/F/TAF
- Part A: Placebo (Placebo Comparator): Participants will receive single dose of placebo matched to lenacapavir on Day 1 followed by B/F/TAF as per standard-care therapy starting on Day 10 through Day 225.
  Interventions: Drug: Placebo; Drug: B/F/TAF
- Part B: TAF 200 mg (Experimental): Participants will receive a single dose of TAF 200 mg on Day 1 followed by B/F/TAF as per standard-care therapy starting on Day 10 through Day 225.
  Interventions: Drug: B/F/TAF; Drug: TAF
- Part B: TAF 600 mg (Experimental): Participants will receive a single dose of TAF 600 mg on Day 1 followed by B/F/TAF as per standard-care therapy starting on Day 10 through Day 225.
  Interventions: Drug: B/F/TAF; Drug: TAF

INTERVENTIONS:
Drug: Lenacapavir — Administered subcutaneously in the abdomen
  Other Names: GS-6207
  Arms: Part A: Lenacapavir 150 mg; Part A: Lenacapavir 20 mg; Part A: Lenacapavir 450 mg; Part A: Lenacapavir 50 mg; Part A: Lenacapavir 750 mg
Drug: Placebo — Administered subcutaneously in the abdomen
  Arms: Part A: Placebo
Drug: B/F/TAF — 50/200/25 mg tablets administered orally once daily
  Other Names: Biktarvy®
Drug: TAF — Tablets administered orally
  Arms: Part B: TAF 200 mg; Part B: TAF 600 mg

SUMMARY:
The primary objectives of this study are:

Part A: To evaluate the short-term antiviral activity of lenacapavir (formerly GS-6207) with respect to the maximum reduction of plasma HIV-1 RNA (log10 copies/mL) from Day 1 through Day 10 compared to placebo in HIV-1 infected adults who are antiretroviral treatment naive or are experienced but capsid inhibitor (CAI) naive.

Part B: To evaluate the short-term antiviral activity of tenofovir alafenamide (TAF) with respect to the maximum reduction of plasma HIV-1 RNA (log10 copies/mL) from Day 1 through Day 10 in HIV-1 infected adult subjects who are antiretroviral treatment naïve or are experienced but without resistance to TAF.

ELIGIBILITY:
Key Inclusion Criteria:

* Plasma HIV-1 RNA ≥ 5,000 copies/mL but ≤ 400,000 copies/mL and CD4+ cell count > 200 cells/mm^3
* Treatment naive or experienced but CAI (for Part A only) and integrase strand transfer inhibitor (INSTI) naïve, and have not received any antiretroviral therapy (ART) within 12 weeks of screening
* Screening genotype report must show sensitivity to B/F/TAF to allow its initiation on Day 10
* Screening genotype report must show sensitivity to at least one agent in either non-nucleoside reverse transcriptase inhibitor (NNRTI) or protease inhibitor (PI) class to allow its use as part of standard of care oral antiretroviral treatment in the future
* Have adequate renal function (estimated glomerular filtration rate ≥ 70 mL/min)
* No clinically significant abnormalities in electrocardiography (ECG) at Screening
* Willing to initiate B/F/TAF on Day 10 after completion of all assessments

Key Exclusion Criteria:

* Pregnant or lactating females

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (12):
- United States (12):
  - Ruane Clinical Research Group, Inc., Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - One Community, Sacramento, California
  - The Lundquist Institute for BioMedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center PA, Orlando, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Be Well Medical Center, Berkley, Michigan
  - AIDS Arms, Inc., DBA Prism Health North Texas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - The Crofoot Research Center, INC (dba Gordon E. Crofoot MD PA), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daar ES, McDonald C, Crofoot G, Ruane P, Sinclair G, Begley R, et al. Dose-response relationship of subcutaneous long-acting HIV capsid inhibitor GS-6207 [Poster]. Presented at: Conference on Retroviruses and Opportunistic Infections; 2020 March 8-11; Boston, MA, USA
- [Result] Daar ES, McDonald C, Crofoot G, Ruane P, Sinclair G, Patel H, et al. Single doses of long acting capsid inhibitor GS-6207 administered by subcutaneous injection are safe and efficacious in people living with HIV [Poster]. Presented at: 17th European AIDS Conference; 2019 November 6-9; Basel, Switzerland.
- [Result] Daar ES, McDonald C, Crofoot G, Ruane P, Sinclair G, Patel H, et al. Safety and antiviral activity over 10 days following a single dose of subcutaneous GS-6207, a first-in-class, long acting HIV capsid inhibitor in people living with HIV [Poster]. Presented at: 10th IAS Conference on HIV Science; 2019 21-24 July; Mexico City, Mexico.
- [Result] Link JO, Rhee MS, Tse WC, Zheng J, Somoza JR, Rowe W, Begley R, Chiu A, Mulato A, Hansen D, Singer E, Tsai LK, Bam RA, Chou CH, Canales E, Brizgys G, Zhang JR, Li J, Graupe M, Morganelli P, Liu Q, Wu Q, Halcomb RL, Saito RD, Schroeder SD, Lazerwith SE, Bondy S, Jin D, Hung M, Novikov N, Liu X, Villasenor AG, Cannizzaro CE, Hu EY, Anderson RL, Appleby TC, Lu B, Mwangi J, Liclican A, Niedziela-Majka A, Papalia GA, Wong MH, Leavitt SA, Xu Y, Koditek D, Stepan GJ, Yu H, Pagratis N, Clancy S, Ahmadyar S, Cai TZ, Sellers S, Wolckenhauer SA, Ling J, Callebaut C, Margot N, Ram RR, Liu YP, Hyland R, Sinclair GI, Ruane PJ, Crofoot GE, McDonald CK, Brainard DM, Lad L, Swaminathan S, Sundquist WI, Sakowicz R, Chester AE, Lee WE, Daar ES, Yant SR, Cihlar T. Clinical targeting of HIV capsid protein with a long-acting small molecule. Nature. 2020 Aug;584(7822):614-618. doi: 10.1038/s41586-020-2443-1. Epub 2020 Jul 1. PMID 32612233
- [Result] Margot N, Ram R, Parvangada P, Martin R, Hyland R, Rhee M, Callebaut C. Lenacapavir resistance analysis in a phase Ib clinical proof-of-concept study [oral]. Presented at: HIV Glasgow; 2020 October 5 - 8; Virtual.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 26 November 2018. The last study visit occurred on 15 June 2020.
Pre-assignment Details: 89 participants were screened.
Groups:
- Part A: Lenacapavir 20 mg: Participants received a single dose of lenacapavir 20 mg subcutaneously in the abdomen on Day 1 followed by bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) as per standard-care therapy started on Day 10 through Day 225.
- Part A: Lenacapavir 50 mg: Participants received a single dose of lenacapavir 50 mg subcutaneously in the abdomen on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
- Part A: Lenacapavir 150 mg: Participants received a single dose of lenacapavir 150 mg subcutaneously in the abdomen on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
- Part A: Lenacapavir 450 mg: Participants received a single dose of lenacapavir 450 mg subcutaneously in the abdomen on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
- Part A: Lenacapavir 750 mg: Participants received a single dose of lenacapavir 750 mg subcutaneously in the abdomen on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
- Part A: Placebo: Participants received a single dose of placebo matched to lenacapavir subcutaneously in the abdomen on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
- Part B: Tenofovir Alafenamide (TAF) 200 mg: Participants received a single oral dose of TAF 200 mg on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
- Part B: TAF 600 mg: Participants received a single oral dose of TAF 600 mg on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
Period: Overall Study
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo | Part B: Tenofovir Alafenamide (TAF) 200 mg | Part B: TAF 600 mg
Started | 6 | 6 | 7 | 6 | 6 | 10 | 7 | 5
Completed | 6 | 6 | 6 | 5 | 5 | 10 | 7 | 5
Not Completed | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Enrolled but not treated | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were randomized/enrolled and received at least 1 dose of study drug.
Groups:
- Part A: Lenacapavir 20 mg: Participants received a single dose of lenacapavir 20 mg subcutaneously in the abdomen on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
- Part B: TAF 200 mg: Participants received a single oral dose of TAF 200 mg on Day 1 followed by B/F/TAF as per standard-care therapy started on Day 10 through Day 225.
- Part B: TAF 600 mg: Participants received a single oral dose of TAF 600 mg on Day 1 followed by B/F/TAF as per standard-care therapy on started on Day 10 through Day 225.
- Total: Total of all reporting groups
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo | Part B: TAF 200 mg | Part B: TAF 600 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10 | 7 | 5 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (4.4) | 36 (14.4) | 39 (11.5) | 36 (15.5) | 37 (17.7) | 29 (9.3) | 29 (8.7) | 40 (8.7) | 34 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 4
  Male | 6 | 6 | 5 | 6 | 3 | 9 | 7 | 5 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 3 | 1 | 5 | 2 | 13
  Not Hispanic or Latino | 5 | 6 | 6 | 5 | 2 | 9 | 2 | 3 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Race: Black | 0 | 2 | 3 | 2 | 1 | 4 | 1 | 0 | 13
  Race: White | 4 | 3 | 2 | 4 | 3 | 5 | 5 | 5 | 31
  Race: Other | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.46 (0.428) | 4.44 (0.328) | 4.48 (0.161) | 4.52 (0.190) | 4.56 (0.305) | 4.50 (0.371) | 4.23 (0.621) | 4.97 (0.439) | 4.50 (0.403)

OUTCOME MEASURES:

1. Primary Outcome: Part A and Part B: Maximum Reduction From Day 1 (Baseline) Through Day 10 in Plasma HIV-1 RNA
Description: Maximum reduction is defined as the minimum of change from baseline in plasma HIV-1 RNA (i.e. smallest change in HIV-RNA from baseline).
Time Frame: Day 1 through Day 10
Population: The Full Analysis Set (FAS) included all participants who were randomized/enrolled and received at least 1 full dose of study drug.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10 | 7 | 5
log10 copies/mL | -1.35 (0.318) | -1.79 (0.476) | -1.76 (0.203) | -2.20 (0.468) | -2.26 (0.662) | -0.17 (0.128) | -0.75 (0.270) | -0.91 (0.294)
Statistical Analysis 1: Comparison: Part A: Lenacapavir 20 mg vs Part A: Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Part A: Lenacapavir 50 mg vs Part A: Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Part A: Lenacapavir 150 mg vs Part A: Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Part A: Lenacapavir 450 mg vs Part A: Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Part A: Lenacapavir 750 mg vs Part A: Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Part A and Part B: Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE could therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs were defined as any AE with an onset date on or after the study drug start date.
Time Frame: Day 1 through 225 days
Population: The Safety Analysis Set included all participants who were randomized/enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10 | 7 | 5
percentage of participants | 83.3 | 100 | 83.3 | 100 | 80 | 70 | 85.7 | 100

3. Secondary Outcome: Part A and Part B: Percentage of Participants Experiencing Treatment Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Day 1 through 225 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10 | 7 | 5
percentage of participants | 83.3 | 83.3 | 100.0 | 66.7 | 100.0 | 80.0 | 100.0 | 80.0

4. Secondary Outcome: Part A and Part B Pharmacokinetic (PK) Parameter: AUCinf of Lenacapavir, TAF and Its Metabolite TFV
Description: AUCinf is defined as area under the concentration versus time curve from time zero to infinity.
Time Frame: Part A: 0 (predose),1,2,4,8,12,24 h postdose on Day 1, anytime on Days 3,4,7,8,9,10,14,29,43,57,85,113,141,169,197,225; Part B: 0 (predose),0.5,1,2,3,4,6,8,10,12,24 and 48 h postdose on Day 1, approximately Day 1 predose time on Days 4,5,6,7,8,9,10
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 7 | 5
h*ng/mL
  Part A: Lenacapavir: number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 0 | 0
  Part A: Lenacapavir | 6564.3 (2562.02) | 9124.1 (4443.03) | 31537.0 (6811.74) | 106041.1 (19939.41) | 181861.0 (73100.91) |  |
  Part B: TAF: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Part B: TAF |  |  |  |  |  | 1270.3 (346.47) | 3556.1 (1396.81)
  Part B: TFV: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Part B: TFV |  |  |  |  |  | 2807.9 (904.23) | 13435.4 (1748.60)

5. Secondary Outcome: Part A and Part B PK Parameter: AUClast of Lenacapavir, TAF and Its Metabolite TFV
Description: AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Error); unit: h*ng/mL
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 7 | 5
h*ng/mL
  Part A: Lenacapavir: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 0 | 0
  Part A: Lenacapavir | 5084.3 (2143.03) | 7524.4 (4140.40) | 28866.4 (8247.37) | 102919.0 (19984.50) | 171173.9 (80524.85) |  |
  Part B: TAF: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Part B: TAF |  |  |  |  |  | 1265.8 (350.75) | 3553.0 (1396.14)
  Part B: TFV: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Part B: TFV |  |  |  |  |  | 2706.7 (877.05) | 12682.5 (1780.31)

6. Secondary Outcome: Part A and Part B PK Parameter: Cmax of Lenacapavir, TAF and Its Metabolite TFV
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 7 | 5
ng/mL
  Part A: Lenacapavir: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 0 | 0
  Part A: Lenacapavir | 3.0 (1.00) | 5.4 (4.00) | 17.1 (7.33) | 60.1 (16.92) | 116.6 (40.38) |  |
  Part B: TAF: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Part B: TAF |  |  |  |  |  | 1919.0 (822.57) | 3934.0 (742.85)
  Part B: TFV: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Part B: TFV |  |  |  |  |  | 93.0 (36.97) | 371.0 (72.76)

7. Secondary Outcome: Part B PK Parameter: AUCinf of TFV-DP Metabolite of TAF
Description: AUCinf is defined as area under the concentration versus time curve from time zero to infinity.
Time Frame: Part B: 0 (predose), 1, 2, 4, 6, 8, 12, 24 and 48 hours post dose on Day 1, approximately Day 1 predose time on Days 4, 5 (if possible), 6 (if possible), 7, 8, 9, 10
Population: The peripheral blood mononuclear cell (PBMC) PK Analysis Set included all participants who are enrolled in Part B of the study, received at least 1 dose of study drug, and had at least 1 nonmissing TFV-DP concentration. Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*uM
Arm/Group | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 4 | 5
h*uM | 599.7 (299.36) | 7981.4 (3852.75)

8. Secondary Outcome: Part B PK Parameter: AUClast of TFV-DP Metabolite of TAF
Description: as for outcome 5
Time Frame: as for outcome 7
Population: Participants in the PBMC PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*uM
Arm/Group | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 5
h*uM | 390.9 (372.31) | 7749.3 (3731.57)

9. Secondary Outcome: Part B PK Parameter: Cmax of TFV-DP Metabolite of TAF
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: as for outcome 7
Population: Participants in the PBMC PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 5
uM | 8.5 (9.94) | 163.0 (118.75)

10. Secondary Outcome: Part A: Percentage of Participants Ever Achieving HIV-1 RNA < 50 Copies/mL by Day 10
Time Frame: Day 10
Population: Participants in the FAS Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 10
percentage of participants | 0 | 16.7 | 0 | 16.7 | 20.0 | 0

11. Secondary Outcome: Part A: Number of Participants Experiencing Any Emergence of Capsid Inhibitor Resistance
Time Frame: Day 10
Population: Participants in the End of Monotherapy Resistance Analysis Population who had received 1 dose of study drug or placebo, regardless of virologic status were analyzed. One participant in 'Part A: Lenacapavir 750 mg' group had assay failure and thus was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 10
Participants | 1 | 1 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part A: Number of Participants Experiencing Any Emergence of Capsid Inhibitor Resistance
Description: Post-Monotherapy Resistance Analysis Population analyzed for this outcome measure included any participant who received at least 1 dose of study drug/placebo, maintained their study drug regimen, & met one of following virologic failure criteria:
  * HIV-1 RNA ≥ 50 copies/mL & < 1 log10 HIV-1 RNA reduction from Day 10 at Day 57 visit, confirmed at a scheduled or unscheduled visit at least 2 weeks following Day 57
  * At any visit following Day 10, after achieving HIV-1 RNA < 50 copies/mL, a rebound in HIV-1 RNA to ≥ 50 copies/mL, which was subsequently confirmed at following scheduled or unscheduled visit; OR At any visit, a > 1 log10 increase in HIV-1 RNA from nadir, which was subsequently confirmed at following scheduled or unscheduled visit;
  * Any participant with HIV-1 RNA ≥ 50 copies/mL at study endpoint or study discontinuation who didn't meet any of criteria above also had protease (PR)/reverse transcriptase (RT), integrase (IN), &capsid (CA) genotyping & phenotyping performed.
Time Frame: Day 10 through Day 225
Population: Participants in the Post-Monotherapy Resistance Analysis Population were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Part B: Number of Participants Experiencing Any Emergence of TAF Resistance
Time Frame: Day 10
Population: Participants in the Post-Monotherapy Resistance Analysis Population were analyzed. One participant in 'Part B: TAF 200 mg' group and one participant in 'Part B: TAF 600 mg' group had assay failure and thus were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

14. Secondary Outcome: Part B: Number of Participants Experiencing Any Emergence of TAF Resistance
Description: TAF Resistance testing was performed for any participant meeting Post-Monotherapy Resistance Analysis Population criteria - it included any participant who received at least 1 dose of study drug/placebo, maintained their study drug regimen, & met one of the following virologic failure criteria:
  * HIV-1 RNA ≥50 copies/mL & < 1 log10 HIV-1 RNA reduction from D10 at the D57 visit, confirmed at scheduled or unscheduled visit at least 2 weeks following D57
  * At any visit following D10, after achieving HIV-1 RNA< 50 copies/mL, a rebound in HIV-1 RNA to ≥50 copies/mL, which was subsequently confirmed at the following scheduled/unscheduled visit; OR At any visit, a > 1 log10 increase in HIV-1 RNA from nadir, which was subsequently confirmed at the following scheduled or unscheduled visit;
  * Any participant with HIV-1 RNA ≥50 copies/mL at study endpoint or study discontinuation who didn't meet any of the criteria above also had PR/RT, IN, and CA genotyping & phenotyping performed.
  D = Day
Time Frame: Day 10 through Day 225
Population: Data was not collected as no participants met the specified Post-Monotherapy Resistance Analysis Population criteria.
Arm/Group | Part B: TAF 200 mg | Part B: TAF 600 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through 225 days
Description: The Safety Analysis Set included all participants who were randomized/enrolled and received at least 1 dose of study drug.
Arm/Group | Part A: Lenacapavir 20 mg | Part A: Lenacapavir 50 mg | Part A: Lenacapavir 150 mg | Part A: Lenacapavir 450 mg | Part A: Lenacapavir 750 mg | Part A: Placebo | Part B: TAF 200 mg | Part B: TAF 600 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/10 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/6 | 0/5 | 1/10 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/6 | 6/6 | 4/5 | 7/10 | 6/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Lenacapavir 20 mg (N=6) | Part A: Lenacapavir 50 mg (N=6) | Part A: Lenacapavir 150 mg (N=6) | Part A: Lenacapavir 450 mg (N=6) | Part A: Lenacapavir 750 mg (N=5) | Part A: Placebo (N=10) | Part B: TAF 200 mg (N=7) | Part B: TAF 600 mg (N=5)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Lenacapavir 20 mg (N=6) | Part A: Lenacapavir 50 mg (N=6) | Part A: Lenacapavir 150 mg (N=6) | Part A: Lenacapavir 450 mg (N=6) | Part A: Lenacapavir 750 mg (N=5) | Part A: Placebo (N=10) | Part B: TAF 200 mg (N=7) | Part B: TAF 600 mg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Anogenital dysplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 3
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injection site bruising (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 1 | 4 | 2 | 2 | 1 | 0 | 0
Injection site induration (General disorders) | 0 | 1 | 3 | 2 | 1 | 1 | 0 | 0
Injection site mass (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Injection site nodule (General disorders) | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 4 | 4 | 4 | 4 | 3 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal chlamydia infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Latent tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 2 | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal gonococcal infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal chlamydia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctitis gonococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syphilis (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 2 | 2 | 3
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Stress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Crystalluria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sterile pyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03739866/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT03739866/SAP_001.pdf